CLINICAL TRIAL: NCT03814135
Title: Randomized, Double-blind, Double-dummy, National, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Two Doses of Hipnos Medication in the Treatment of Adults With Insomnia
Brief Title: Efficacy and Safety of Two Doses of Hipnos in the Treatment of Adults With Insomnia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0518 - HIPNOS
Record Dates: First submitted 2019-01-22; First posted 2019-01-23 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Insomnia
Keywords: insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Duble-blind and double-dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIPNOS 3 (Experimental): The study is double-dummy. Thus, the patient will take 2 tablets, as follow:
  1 tablet Hipnos 3 and 1 placebo tablet, oral, once a day.
  Interventions: Drug: Hipnos 3; Other: Hipnos 5 Placebo
- HIPNOS 5 (Experimental): The study is double-dummy. Thus, the patient will take 2 tablets, as follow:
  1 tablet Hipnos 5 and 1 placebo tablet, oral, once a day.
  Interventions: Drug: Hipnos 5; Other: Hipnos 3 Placebo
- HIPNOS Placebo (Placebo Comparator): The study is double-dummy. Thus, the patient will take 2 tablet of placebo, oral, once a day.
  Interventions: Other: Hipnos 5 Placebo; Other: Hipnos 3 Placebo

INTERVENTIONS:
Drug: Hipnos 3 — 1 tablet, oral, once a day.
  Other Names: EMS tablet
  Arms: HIPNOS 3
Drug: Hipnos 5 — 1 tablet, oral, once a day.
  Other Names: EMS tablet
  Arms: HIPNOS 5
Other: Hipnos 5 Placebo — 1 tablet, oral, once a day.
  Other Names: Placebo
  Arms: HIPNOS 3; HIPNOS Placebo
Other: Hipnos 3 Placebo — 1 tablet, oral, once a day.
  Other Names: Placebo
  Arms: HIPNOS 5; HIPNOS Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of three doses of Hipnos medication in adults with insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 50 years or more;
* Diagnosis of insomnia disorder according to criteria defined by the DSM-V;
* Sleep latency ≥ 20 minutes obtained through polysomnography performed prior to the randomization visit.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Known hypersensitivity to the formula components used during the clinical trial;
* Decompensated diabetes mellitus, hypothyroidism or hyperthyroidism;
* History of hepatic impairment;
* Current smoking;
* Pregnancy or risk of pregnancy and lactating patients;
* History of sleep-disordered breathing, sleep disorders associated with changes in circadian rhythm and severe neurological and psychiatric disorders;
* Diagnosis of clinical diseases that interfere with sleep;
* Participants who have used psychostimulant medications, antidepressants and/ or antipsychotic with sedative effects and/or antiepileptic;
* Participation in clinical trial in the year prior to this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change in sleep latency time, obtained through polysomnography, performed before and at the end of treatment. | 4 weeks

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 5 weeks